CLINICAL TRIAL: NCT02273596
Title: A Phase 2, Multi-centre, Open-label, Study to Evaluate the Efficacy and Safety of WTX101 Administered for 24 Weeks in Newly Diagnosed Wilson Disease Patients Aged 18 and Older With an Extension Phase of 36 Months
Brief Title: Efficacy and Safety Study of WTX101 (ALXN1840) in Adult Wilson Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WTX101-201
Record Dates: First submitted 2014-10-20; First posted 2014-10-24 (Estimated); Results first posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALXN1840 (Experimental): Treatment Period: ALXN1840 at individualized doses ranging from 15 to 60 milligram (mg) per day. Dose increases or dose reductions were dependent on the individual NCC concentrations adjusted for Mo plasma concentration. ALXN1840 may have been administered every other day, once daily, or twice daily, depending on individualized dosing regimen, for 24 weeks.
  Extension Period: Participants continued the same ALXN1840 daily dose maintained at Week 24 of the Treatment Period and the same dosing regimen. During the Extension Period, no up-titration was made unless NCC concentrations adjusted for Mo plasma concentration did not remain stable within (or below) the reference range. ALXN1840 could have been received for up to 36 months in the Extension Period.
  Interventions: Drug: ALXN1840

INTERVENTIONS:
Drug: ALXN1840 — Individualized oral doses of ALXN1840.
  Other Names: WTX101

SUMMARY:
The main purpose of the study was to evaluate the efficacy of ALXN1840 (formerly WTX101) for 24 weeks on non-ceruloplasmin-bound copper (NCC) concentrations adjusted for molybdenum plasma concentration in participants newly diagnosed with Wilson Disease (WD) who were aged 18 and older and who had NCC concentrations within or above the reference range at the time of enrollment in the study. The study consisted of a 24-week Treatment Period, followed by a planned 36-month Extension Period.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to comply with study procedures, restrictions, and requirements, as judged by the Investigator.
* Newly established diagnosis of WD by Leipzig-Score ≥ 4 documented by testing as outlined in 2012 European Association for the Study of the Liver Wilson Disease Clinical Practice Guidelines.
* NCC levels within or above the normal reference range (0.8 to 2.3 micromole).
* Willing to undergo 48 hour washout from current WD treatment

Exclusion Criteria:

* Treatment for greater than 24 months for WD with chelation therapy (for example, penicillamine, trientine hydrochloride) or zinc therapy.
* Decompensated hepatic cirrhosis.
* Model for End-Stage Liver Disease score > 11.
* Modified Nazer score > 6.
* Gastrointestinal bleed within past 6 months.
* Alanine aminotransferase > 5 x upper limit of normal.
* Marked neurological disease requiring either nasogastric feeding or intensive in-patient medical care.
* Severe anemia with a hemoglobin < 9 grams/deciliter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2016-10-27 (Actual); Study Completion 2018-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Swenson, MD, PhD, Study Director — Alexion Pharmaceuticals, Inc.
Locations (9):
- United States (4):
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, New Haven, Connecticut
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Ann Arbor, Michigan
- Clinical Trial Site, Vienna, Austria
- Clinical Trial Site, Heidelberg, Germany
- Clinical Trial Site, Warsaw, Poland
- United Kingdom (2):
  - Clinical Trial Site, Guildford, Surrey
  - Clinical Trial Site, Birmingham

REFERENCES:
- [Result] Weiss KH, Askari FK, Czlonkowska A, Ferenci P, Bronstein JM, Bega D, Ala A, Nicholl D, Flint S, Olsson L, Plitz T, Bjartmar C, Schilsky ML. Bis-choline tetrathiomolybdate in patients with Wilson's disease: an open-label, multicentre, phase 2 study. Lancet Gastroenterol Hepatol. 2017 Dec;2(12):869-876. doi: 10.1016/S2468-1253(17)30293-5. Epub 2017 Oct 5. PMID 28988934

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants meeting all inclusion and no exclusion criteria were enrolled into the study and studied as outpatients. Participants enrolled as pre-treated with other de-coppering agents were required to undergo a 48-hour washout from their previous Wilson Disease (WD) treatment just prior to initiation of study treatment. Participants who completed the 24-week treatment period and had favorable safety profiles and WD control were offered the opportunity to participate in the Extension Period.
Groups:
- ALXN1840: Treatment Period: ALXN1840 at individualized doses ranging from 15 to 60 milligrams (mg) per day. Dose increases or dose reductions were dependent on the individual non-ceruloplasmin-bound copper (NCC) concentrations adjusted for molybdenum (Mo) plasma concentration. ALXN1840 may have been administered every other day, once daily, or twice daily, depending on individualized dosing regimen, for 24 weeks.
  Extension Period: Participants continued the same ALXN1840 daily dose maintained at Week 24 of the Treatment Period and the same dosing regimen. During the Extension Period, no up-titration was made unless NCC concentrations adjusted for Mo plasma concentration did not remain stable within (or below) the reference range.
Period: 24-Week Treatment Period
Arm/Group | ALXN1840
Started | 29
Received at Least 1 Dose of Study Drug (One participant was enrolled but not treated) | 28
Completed | 22
Not Completed | 7
Not completed — Adverse Event | 3
Not completed — Withdrawal by Participant Prior to First Dose | 1
Not completed — Participant was unable to Come | 1
Not completed — Physician Decision | 1
Not completed — Protocol Deviation | 1
Period: Extension Period
Arm/Group | ALXN1840
Started | 22
Received at Least 1 Dose of Study Drug | 22
Completed (19 participants who completed the 24-week treatment period were considered to have discontinued Study WTX101-201 to enter Study WTX101-301 (NCT03403205)) | 0
Not Completed | 22
Not completed — Continued into Study WTX101-301 extension (NCT03403205). | 19
Not completed — Participant Withdrew for Personal Reasons | 1
Not completed — Lost to Follow-up | 1
Not completed — Protocol Deviation | 1

BASELINE CHARACTERISTICS:
Population: Participants who were enrolled and received at least 1 dose of study drug.
Groups:
- ALXN1840: Treatment Period: ALXN1840 at individualized doses ranging from 15 to 60 mg per day. Dose increases or dose reductions were dependent on the individual NCC concentrations adjusted for Mo plasma concentration. ALXN1840 may have been administered every other day, once daily, or twice daily, depending on individualized dosing regimen, for 24 weeks.
  Extension Period: Participants continued the same ALXN1840 daily dose maintained at Week 24 of the Treatment Period and the same dosing regimen. During the Extension Period, no up-titration was made unless NCC concentrations adjusted for Mo plasma concentration did not remain stable within (or below) the reference range.
Arm/Group | ALXN1840
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Participants With Normalized Concentrations Of NCC
Description: Normalized concentrations of NCC was defined as who achieving or maintaining normalized levels of NCC (0.8 to 2.3 micromole [μmol]l/liter [L]]) adjusted for Mo plasma concentration or reaching a reduction of at least 25% in NCC corrected for Mo if above the normal reference range at the time of enrollment. NCC was calculated by subtracting the amount of copper (Cu) bound to ceruloplasmin (CP) from the total plasma Cu concentration. Post-baseline NCC values were adjusted (corrected) to account for Cu bound in tripartite complexes with ALXN1840 and albumin. Descriptive statistics are reported.
Time Frame: Week 24
Population: Participants who were enrolled and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- ALXN1840: Treatment Period: ALXN1840 at individualized doses ranging from 15 to 60 mg per day. Dose increases or dose reductions were dependent on the individual NCC concentrations adjusted for Mo plasma concentration. ALXN1840 may have been administered every other day, once daily, or twice daily, depending on individualized dosing regimen, for 24 weeks.
Arm/Group | ALXN1840
Number analyzed (Participants) | 28
percentage of participants | 85.7 [70.8 to 97.6]

2. Secondary Outcome: Change From Baseline In NCC Concentrations Adjusted For Mo Plasma Concentration At Week 24
Description: The change from Baseline in NCC adjusted for Mo plasma concentration over 24 weeks were analyzed and descriptive statistics are reported. Change from Baseline = (Week 24 NCC concentrations adjusted for Mo plasma concentration) - (Baseline NCC concentrations). Least square means and their 95% confidence intervals (CIs) were calculated using a restricted maximum likelihood (REML)-based mixed model for repeated measures (MMRM) with fixed effects for Baseline, cohort, visit, Baseline-by-visit, and cohort-by-visit interaction.
Time Frame: Baseline, Week 24
Population: Participants who were enrolled and received at least 1 dose of study drug and had analyzable data at the specified timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: μmol/L
Arm/Group | ALXN1840
Number analyzed (Participants) | 21
μmol/L | -2.56 [-3.13 to -1.98]

3. Secondary Outcome: Time To Normalization Of NCC Adjusted For Mo Plasma Concentration In Participants With Elevated Baseline NCC
Description: For time to normalization of NCC adjusted for Mo plasma concentration, a Kaplan-Meier approach was used where participants not normalized were censored at the latest observed time point. To achieve a normalized NCC concentration, participants must have demonstrated 2 consecutive measures within the normal range (0.8 to 2.3 μmol/L). Analyses includes all data up to the last assessment in the extension period for participants who reached the event of normalization of NCC corrected concentrations. Last Assessment is a summary of the last available post-baseline result for each participant. Analyses includes all data up to the last assessment in the extension period; up to Week 176.
Time Frame: Up to last assessment (up to Week 176)
Population: This analysis was only performed on the subset of participants with elevated Baseline NCC who reached the event of normalization of NCC corrected concentrations.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ALXN1840
Number analyzed (Participants) | 16
days | 147.5 [37.0 to 211.0]

4. Secondary Outcome: Change From Baseline In Neurological Status Using The Unified Wilson's Disease Rating Scale (UWDRS) (Neurological Subscore; Part I) At Week 24
Description: The UWDRS is a clinical rating scale designed to evaluate the neurological manifestations of WD. Change from Baseline in the UWDRS I for consciousness is presented.
  * UWDRS I: range 0 to 3, maximum score of 3
  * UWDRS I was assessed by a Neurologist
  * Change from Baseline was calculated as: Week 24 score - Baseline score. A decrease in score from Baseline is indicative of both an improvement in condition and a better outcome.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ALXN1840
Number analyzed (Participants) | 22
score on a scale | 0.0 (0.0)

5. Secondary Outcome: Change From Baseline In Neurological Status Using The UWDRS (Neurological Subscore; Parts II, III, And Total Score) At Week 24
Description: The UWDRS is a clinical rating scale designed to evaluate the neurological manifestations of WD. UWDRS comprises 3 parts: UWDRS I (consciousness), UWDRS II (disability), and UWDRS III (neurological status). Change from Baseline in the UWDRS II, III, and total score are presented.
  * UWDRS I: range 0 to 3, maximum score of 3
  * UWDRS II: range 0 to 40, maximum score of 40
  * UWDRS III: range 0 to 175, maximum score of 175
  * UWDRS total score: sum of the UWDRS I, II, and III: range 0 to 218, maximum score of 218
  * UWDRS I and III were assessed by a neurologist, while UWDRS II was reported by the participant or caregiver.
  * Change from Baseline was calculated as: Week 24 score - Baseline score. Least square means and their 95% CIs were calculated using a REML-based MMRM with fixed effects for Baseline, cohort, visit, Baseline-by-visit, and cohort-by-visit interaction. A decrease in score from Baseline is indicative of an improvement in condition and a better outcome.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ALXN1840
Number analyzed (Participants) | 22
score on a scale
  UWDRS Part II | -2.5 [-4.6 to -0.4]
  UWDRS Part III | -5.75 [-10.74 to -0.77]
  Total Score | -8.23 [-15.42 to -1.04]

6. Secondary Outcome: Change From Baseline In Psychiatric Status Dimension Using Mini International Neuropsychiatric Interview (M.I.N.I.) Tracking Standardized Scores At Week 24
Description: The M.I.N.I. is a short structured diagnostic interview for the Diagnostic and Statistical Manual of Mental Disorders IV and the 10th revision of the International Statistical Classification of Diseases and Related Health Problems. It was used to "track" the severity of symptoms by using a combination of questions in 16 Psychiatric Status dimensions that are summarized using a single standardized score for each dimension, ranging from 0 (interpreted as "did not occur at all") to 4 (interpreted as "occurred extremely often"). The standardized score is an average of these responses.
  Change from Baseline = Week 24 standardized score - Baseline standardized score. Least square means and 95% CIs were calculated using an REML-based MMRM with fixed effects for Baseline, cohort, visit, Baseline-by-visit, and cohort-by-visit interaction.
  Decrease from Baseline (a lower score) is indicative of a decrease in symptoms and a better outcome.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ALXN1840
Number analyzed (Participants) | 23
score on a scale
  Major Depressive Episode Standardized: number analyzed (Participants) | 22
  Major Depressive Episode Standardized | -0.39 [-0.62 to -0.16]
  Suicidality Tracking Scale Standardized | -0.07 [-0.09 to -0.04]
  Manic/Hypomanic Episode Standardized: number analyzed (Participants) | 21
  Manic/Hypomanic Episode Standardized | -0.09 [-0.23 to 0.05]
  Panic Disorder Standardized | -0.28 [-0.35 to -0.21]
  Agoraphobia Standardized: number analyzed (Participants) | 22
  Agoraphobia Standardized | -0.58 [-0.70 to -0.46]
  Social Anxiety Disorder Standardized: number analyzed (Participants) | 22
  Social Anxiety Disorder Standardized | -0.35 [-0.52 to -0.18]
  Obsessive Compulsive Disorder Standardized | -0.04 [-0.14 to 0.05]
  Post Traumatic Stress Disorder Standardized: number analyzed (Participants) | 22
  Post Traumatic Stress Disorder Standardized | -0.24 [-0.35 to -0.13]
  Alcohol Use Disorder Standardized: number analyzed (Participants) | 22
  Alcohol Use Disorder Standardized | 0.00 [-0.03 to 0.03]
  Substance Use Disorder Standardized | -0.02 [-0.10 to 0.05]
  Psychotic Disorders Standardized: number analyzed (Participants) | 22
  Psychotic Disorders Standardized | 0.00 [-0.06 to 0.07]
  Anorexia Nervosa Standardized | 0.04 [-0.07 to 0.15]
  Bulimia Nervosa Standardized | 0.0 [-0.12 to 0.13]
  Binge Eating Disorder Standardized: number analyzed (Participants) | 22
  Binge Eating Disorder Standardized | 0.04 [-0.06 to 0.14]
  Generalized Anxiety Disorder Standardized | -0.37 [-0.59 to -0.16]
  Antisocial Personality Disorder Standardized: number analyzed (Participants) | 20
  Antisocial Personality Disorder Standardized | -0.06 [-0.12 to 0.00]

7. Secondary Outcome: Clinical Global Impression-Improvement Scale (CGI-I) At Week 24
Description: The CGI-I is a 7-point scale where the clinician assessed how much participant's illness improved or worsened relative to a Baseline state at the beginning of the intervention and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
  Change from Baseline = Week 24 score - Baseline score. An increase in CGI-I score indicates improvement.
Time Frame: Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ALXN1840
Number analyzed (Participants) | 22
score on a scale | -0.8 [-1.4 to -0.3]

8. Secondary Outcome: Change From Baseline In Clinical Global Impression Severity Scale (CGI-S) At Week 24
Description: The CGI-S is a 7-point scale where the investigator rated severity of participant's illness at the time of assessment, relative to the investigator's past experience with participants who have the same diagnosis. Considering total clinical experience, a participant was assessed on severity of illness at time of rating as: 1, normal, not at all ill; 2, borderline ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  Change from Baseline = Week 24 score - Baseline score. Decrease in CGI-S score and increase indicates improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ALXN1840
Number analyzed (Participants) | 8
score on a scale | -0.9 [-1.7 to 0.0]

9. Secondary Outcome: Change From Baseline In Quality Of Life (QoL)/Patient Reported Outcome (PRO) Assessed By The European Quality Of Life 5 Dimensions (EQ-5D) Visual Analogue Scale (VAS) At Week 24
Description: The EQ-5D VAS records the participant's self-rated health as indicated on a scale from 0 to 100 with 0 being "the worst health you can imagine" and 100 being "the best health you can imagine, with higher scores for a higher quality of life. Change from Baseline = Week 24 score - Baseline score. An increase in score indicates improvement.
  The least-square means and their 95% CIs were calculated using a REML-based MMRM with fixed effects for Baseline, cohort, visit, Baseline-by-visit, and cohort-by-visit interaction.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- ALXN1840: Treatment Period: ALXN1840 at individualized doses ranging from 15 to 60 milligram (mg) per day. Dose increases or dose reductions were dependent on the individual NCC concentrations adjusted for Mo plasma concentration. ALXN1840 may have been administered every other day, once daily, or twice daily, depending on individualized dosing regimen, for 24 weeks.
Arm/Group | ALXN1840
Number analyzed (Participants) | 23
score on a scale | 11.3 [5.1 to 17.6]

10. Secondary Outcome: Change From Baseline In Quality Of Life (QoL)/Patient Reported Outcome (PRO) Assessed By The EQ-5D Descriptive System UK Health Index Scores At Week 24
Description: The EQ-5D-5L Descriptive System provides a simple descriptive profile and a single index value for health status (United Kingdom [UK] Health Index Score). The EQ-5D-5L consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each of which can have 1 of 5 responses that represent 5 levels of severity (no problems, slight problems, moderate problems, severe problems, extreme problems). The participant was asked to indicate his/her health state for each of the 5 dimensions. The 5-item index score was transformed into a utility score between 0 (worst health state) and 1 (best health state).
  Change from Baseline = Week 24 index score - Baseline index score. An increase in score indicates improvement.
  The least square means and their 95% CIs were calculated using a REML-based MMRM with fixed effects for Baseline, cohort, visit, Baseline-by-visit, and cohort-by-visit interaction.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: EQ-5D-5L index score
Arm/Group | ALXN1840
Number analyzed (Participants) | 23
EQ-5D-5L index score | 0.0439 [-0.0341 to 0.1219]

11. Secondary Outcome: QoL/PRO Assessed By The 8-Item Medication Adherence Scale (MMAS-8) At Week 24
Description: The MMAS-8 is a scale used to evaluate adherence to medication. The MMAS-8 consists of 8 questions with a sum score ranging between 0 and 8 points, with 8 being the maximum adherence to medication. Mean adherence to medication is presented.
Time Frame: Week 24
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ALXN1840
Number analyzed (Participants) | 23
score on a scale | 7.59 [7.29 to 7.88]

12. Secondary Outcome: QoL/PRO Assessed By The Treatment Satisfaction Questionnaire For Medication (TSQM-9) At Week 24
Description: The TSQM-9 was used to assess the overall level of satisfaction or dissatisfaction with medication participants were taking. This composite scale is comprised of 2 items on the TSQM-9 survey:
  How satisfied are you that good things about this medication outweigh the bad things? Taking all things into account, how satisfied or dissatisfied are you with this medication? The TSQM-9 domain scores (effectiveness score, convenience score, global satisfaction score) range from 0 to 100 with higher scores representing greater satisfaction for the domain.
Time Frame: Week 24
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ALXN1840
Number analyzed (Participants) | 23
score on a scale
  Effectiveness | 69.81 [58.90 to 80.72]
  Convenience | 83.57 [77.62 to 89.53]
  Global Satisfaction | 75.47 [62.77 to 88.16]

13. Secondary Outcome: Change From Baseline In Hepatic Laboratory Measure Alanine Aminotransferase (ALT) At Week 24
Description: Assessed by laboratory measurements. Change from Baseline = Week 24 ALT level - Baseline ALT level.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ALXN1840
Number analyzed (Participants) | 23
U/L | -2.0 (23.71)

14. Secondary Outcome: Change From Baseline In Hepatic Laboratory Measure Aspartate Aminotransferase (AST) At Week 24
Description: Assessed by laboratory measurements. Change from Baseline = Week 24 AST level - Baseline AST level.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ALXN1840
Number analyzed (Participants) | 23
U/L | -10.3 (28.18)

15. Secondary Outcome: Change From Baseline In Hepatic Laboratory Measure International Normalized Ratio (INR) At Week 24
Description: Assessed by laboratory measurements. Change from Baseline = Week 24 INR - Baseline INR.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ALXN1840
Number analyzed (Participants) | 22
ratio | -0.05 (0.148)

16. Secondary Outcome: Change From Baseline In Hepatic Laboratory Measure Bilirubin At Week 24
Description: Assessed by laboratory measurements. Change from Baseline = Week 24 bilirubin level - Baseline bilirubin level.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | ALXN1840
Number analyzed (Participants) | 23
μmol/L | -0.7 (4.30)

17. Secondary Outcome: Change From Baseline In Exchangeable Cu At Week 24
Description: Assessed by laboratory measurements. Change from Baseline = Week 24 Exchangeable Cu level - Baseline Exchangeable Cu level.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ALXN1840
Number analyzed (Participants) | 22
ng/mL | -25.1 (56.64)

18. Secondary Outcome: Change From Baseline In Speciation Profiling (Mo, Cu, And Protein Complex Profiling Using Size Exclusion Chromatography) At Week 24
Description: Due to low chromatographic resolution of data, quantitative analysis for speciation profiling, as had been planned in the protocol, was not feasible.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Arm/Group | ALXN1840
Number analyzed (Participants) | 0

19. Secondary Outcome: Change From Baseline In 24-Hour Urinary Mo And Cu At Week 24
Description: Assessed by laboratory measurements. Change from Baseline = Week 24 (24-hour) urinary Mo or Cu level - Baseline 24-hour urinary Mo or Cu level.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: μg/day
Arm/Group | ALXN1840
Number analyzed (Participants) | 20
μg/day
  Mo | 1561.1 [1093.8 to 2028.4]
  Cu | -28.1 [-107.1 to 51.0]

20. Secondary Outcome: Pharmacokinetics (PK): Area Under The Curve From Time 0 to 24 (AUC0-24) Of Plasma Total Mo
Description: PK blood sampling occurred on Day 1, Week 12, and Week 24 at the following serial PK sampling time-points: 0, 1, 2, 3, 4, 5, 6, 8, and 12 (10 to 12) hours post-dose.
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, and 12 (10 to 12) hours post-dose on Day 1, Week 12, and Week 24
Population: Participants who were enrolled and received at least 1 dose of study drug and had any Baseline and post-Baseline measurable concentration data reported.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- ALXN1840 Every Other Day: ALXN1840 administered at 15 mg every other day.
- ALXN1840 15 mg Daily: ALXN1840 administered at 15 mg per day.
- ALXN1840 30 mg Daily: ALXN1840 administered at 30 mg per day.
- ALXN1840 60 mg Daily: ALXN1840 administered at 60 mg per day (or 30 mg twice daily).
Arm/Group | ALXN1840 Every Other Day | ALXN1840 15 mg Daily | ALXN1840 30 mg Daily | ALXN1840 60 mg Daily
Number analyzed (Participants) | 1 | 4 | 16 | 6
h*ng/mL
  Day 1: number analyzed (Participants) | 0 | 3 | 16 | 2
  Day 1 |  | 2872.6 (943.4) | 4796.7 (3464.8) | 3138.7 (3090.3)
  Week 12: number analyzed (Participants) | 0 | 4 | 13 | 6
  Week 12 |  | 7873.6 (3361.1) | 8836.9 (2675.9) | 11342.5 (4706.7)
  Week 24: number analyzed (Participants) | 1 | 3 | 8 | 5
  Week 24 | 5668.7 (NA) — Not available due to small sample size | 4593.6 (1260.0) | 7884.3 (3157.2) | 8890.2 (5801.6)

21. Secondary Outcome: PK: Maximum Concentration (Cmax) Of Plasma Total Mo
Description: as for outcome 20
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, and 12 (10 to 12) hours post-dose on Day 1, Week 12, and Week 24
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ALXN1840 Every Other Day | ALXN1840 15 mg Daily | ALXN1840 30 mg Daily | ALXN1840 60 mg Daily
Number analyzed (Participants) | 1 | 6 | 19 | 7
ng/mL
  Day 1: number analyzed (Participants) | 0 | 6 | 19 | 3
  Day 1 |  | 202.7 (114.5) | 304.8 (202.9) | 167.6 (144.6)
  Week 12: number analyzed (Participants) | 0 | 6 | 14 | 6
  Week 12 |  | 393.0 (177.3) | 488.8 (165.5) | 607.3 (257.3)
  Week 24: number analyzed (Participants) | 1 | 4 | 10 | 7
  Week 24 | 364.0 (NA) — Not available due to small sample size | 359.0 (163.7) | 447.7 (200.4) | 489.9 (293.4)

22. Secondary Outcome: Extension Period: Percentage Of Participants With Normalized Concentrations Of NCC
Description: Normalized concentrations of NCC was defined as who achieving or maintaining normalized levels of NCC (0.8-2.3 μM) adjusted for Mo plasma concentration or reaching a reduction of at least 25% in NCC corrected for Mo if above the normal reference range at the time of enrollment. NCC was calculated by subtracting the amount of Cu bound to Cp from the total plasma Cu concentration. Post-baseline NCC values were adjusted (corrected) to account for Cu bound in tripartite complexes with ALXN1840 and albumin. Last Assessment is a summary of the last available post-baseline result for each participant. Analyses includes all data up to the last assessment in the extension period; up to Week 176.
Time Frame: Up to last assessment (up to Week 176)
Population: Participants who were enrolled and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ALXN1840
Number analyzed (Participants) | 28
percentage of participants | 92.9 [81.0 to 99.9]

23. Secondary Outcome: Extension Period: Change From Baseline In NCC Levels Adjusted For Mo Plasma Concentration
Description: The change from Baseline in NCC adjusted for Mo plasma concentration over 176 weeks were analyzed. Last Assessment is a summary of the last available post-baseline result for each participant. Analyses includes all data up to the last assessment in the extension period, up to Week 176. Change from Baseline = (Last assessment [up to Week 176] NCC concentrations adjusted for Mo plasma concentration) - (Baseline NCC concentrations). Least square means and their 95% CIs were calculated using an REML-based MMRM with fixed effects for Baseline, cohort, visit, Baseline-by-visit, and cohort-by-visit interaction.
Time Frame: Baseline, last assessment (up to Week 176)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: μmol/L
Arm/Group | ALXN1840
Number analyzed (Participants) | 25
μmol/L | -2.92 [-3.45 to -2.39]

ADVERSE EVENTS:
Time Frame: Day 1 after dosing up to last assessment (up to Week 176), mean duration of treatment of 693.1 days
Arm/Group | ALXN1840
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 11/28
Other Adverse Events (participants affected / at risk) | 26/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALXN1840 (N=28)
Agranulocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Hepato-lenticular degeneration (Congenital, familial and genetic disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gait disturbance (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neurological decompensation (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Abnormal behaviour (Psychiatric disorders) | 1
Adjustment disorder (Psychiatric disorders) | 1
Affective disorder (Psychiatric disorders) | 1
Mania (Psychiatric disorders) | 1
Personality disorder (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALXN1840 (N=28)
Leukopenia (Blood and lymphatic system disorders) | 3
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 6
Urinary tract infection (Infections and infestations) | 8
Sinusitis (Infections and infestations) | 3
Influenza (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 9
Gamma-glutamyltransferase increased (Investigations) | 8
Hepatic enzyme increased (Investigations) | 6
Blood alkaline phosphatase increased (Investigations) | 3
Blood creatine phosphokinase increased (Investigations) | 2
Liver function test increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 6
Tremor (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Sleep disorder (Psychiatric disorders) | 3
Depressed mood (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
Due to low chromatographic resolution of data, quantitative analysis for speciation profiling, as had been planned in the protocol, was not feasible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes